CLINICAL TRIAL: NCT04423770
Title: COVID-19 Related Health and Infection Control Practices Among Dentists
Status: Completed | Type: Observational
Sponsor: American Dental Association (Other)
Responsible Party: Principal Investigator, Cameron Estrich, Health Research Analyst, American Dental Association
Other Study IDs: 20-08
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: SARS-CoV-2; COVID-19; survey; dentistry; infection control
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- U.S. dentists: Dentists in the United States
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention; this is a purely observational study

SUMMARY:
As dentists begin reopening their practices during a global pandemic, the risk of COVID-19 infection that dentists face in providing dental care remains unknown. Estimating the occupational risk of COVID-19, and producing evidence on the types of infection control practices and dental practices that may affect COVID-19 risk, is therefore imperative. The goal of the proposed study is to understand U.S.-based dentists' health and dental-practice reactions to COVID-19. To estimate this, U.S-based dentists will be surveyed monthly. These findings could be used to describe the prevalence and incidence of COVID-19 among dentists, determine what infection control steps dentists take over time, and estimate whether infection control adherence in dental practice is related to COVID-19 incidence.

ELIGIBILITY:
Inclusion Criteria:

* Primary dental practice is in United States
* 18 years of age or older
* Dentist

Exclusion Criteria:

•Answered "no" to ADA survey sent May 2020 that read "As part of ongoing efforts to monitor the effect of COVID-19 on the dental team, the ADA is interested in collecting data related to infection rates. Would you also be willing to participate in a separate, longitudinal study that would require you to report whether you or your staff have exhibited symptoms of COVID-19, and whether you have been tested or diagnosed? The study would be anonymous and under IRB protocols."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dentists in the United States
Sampling Method: Non-Probability Sample
Enrollment: 2196 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
COVID-19 probable or confirmed case | 18 months
  COVID-19 case as confirmed by clinician and/or detection of SARS-CoV-2 RNA or a specific antigen in a clinical specimen

SECONDARY OUTCOMES:
Anxiety | 12 months
  Assessed using the Patient Health Questionnaire for Depression and Anxiety (PHQ-4). Two items scored 0 to 3 (total score of 0-6), with higher numbers indicating greater anxiety.
Depression | 12 months
  Assessed using the Patient Health Questionnaire for Depression and Anxiety (PHQ-4). Two items scored 0 to 3 (total score of 0-6), with higher numbers indicating greater depressive symptoms.
Dental practice infection control efforts | 12 months
  Self-reports of infection control efforts in the respondents' primary dental practices
Dentists' use of personal protective equipment | 12 months
  Self-reports of personal protective equipment use

CONTACTS AND LOCATIONS:
Overall Officials: Cameron G Estrich, MPH, PhD, Principal Investigator — American Dental Association Science and Research Institute
Locations (1):
- American Dental Association, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eldridge LA, Estrich CG, Gurenlian JR, Battrell A, Lynch A, Vujicic M, Morrissey R, Dershewitz S, Geisinger ML, Araujo MWB. US dental health care workers' mental health during the COVID-19 pandemic. J Am Dent Assoc. 2022 Aug;153(8):740-749. doi: 10.1016/j.adaj.2022.02.011. PMID 35902154
- [Derived] Estrich CG, Mikkelsen M, Morrissey R, Geisinger ML, Ioannidou E, Vujicic M, Araujo MWB. Estimating COVID-19 prevalence and infection control practices among US dentists. J Am Dent Assoc. 2020 Nov;151(11):815-824. doi: 10.1016/j.adaj.2020.09.005. PMID 33071007